CLINICAL TRIAL: NCT05478005
Title: Comparison of Function and Pain Intensity in the Acute Stage Following Total Knee Replacement, Between Different Methods of Post-surgical Pain Relief
Brief Title: Function and Pain Following Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Michal Elboim, Full-time lecturer and faculty member in the Physical Therapy Department at the University of Haifa (UOH), University of Haifa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHaifa-MEGK
Record Dates: First submitted 2022-07-04; First posted 2022-07-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Knee Arthropathy; Post Operative Pain; Pain, Postoperative
Keywords: post operative pain; total knee replacement; total knee arthroplasty; pain; post operative function; nerve block; intra-articular block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who was blinded to the treatment group allocation and who was not involved in the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Femoral nerve block (Experimental): Patients undergoing total knee arthroplasty received a single-shot femoral nerve block during the surgical procedure.
  Interventions: Procedure: Femoral nerve block
- Intra-articular block (Experimental): Patients undergoing total knee arthroplasty received a intra-articular block during the surgical procedure.
  Interventions: Procedure: Intra-articular block
- Control group (No Intervention): Patients undergoing total knee arthroplasty and didn't receive pain block.

INTERVENTIONS:
Procedure: Femoral nerve block — Patients who receive a femoral nerve block during surgery, fill out a questionnaire and undergo a muscle strength test before surgery, undergo functional tests, a muscle strength test and are asked about pain intensity after surgery.
  Arms: Femoral nerve block
Procedure: Intra-articular block — Patients who receive an intra-articular block at the time of surgery, fill out a questionnaire and undergo a muscle strength test before surgery, undergo functional tests, a muscle strength test and are asked about pain intensity after surgery.
  Arms: Intra-articular block

SUMMARY:
The goal of this interventional study is to compare pain management techniques (femoral nerve block, intra-articular block, none) in TKA patients. The main questions it aims to answer are:

* Are there differences in postoperative outcomes?
* Does preoperative quadriceps muscle strength predict early functional ability? Participants underwent TKA and assessments. Researchers compared pain management techniques to assess effects on postoperative outcomes and identified the importance of preoperative quadriceps muscle strength as a predictor of early functional ability. Further research is required to refine postoperative pain management strategies.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is a frequently undertaken elective orthopedic intervention for severe knee osteoarthritis, frequently yielding postoperative discomfort and complications. Peripheral nerve blocks, notably femoral nerve blocks, are commonly utilized for analgesia but may transiently impede motor nerve function, weakening the quadriceps muscle. Intra-articular blocks offer a potential alternative to mitigate motor impairment. However, there exists a dearth of information regarding the comparative effectiveness of these methods with respect to short-term functional outcomes in the immediate postoperative phase following TKA.

Objectives: This study assesses functional outcomes, pain, quadriceps strength after TKA with femoral nerve block, intra-articular block, and a control group. It identifies predictors of postoperative functional ability.

Methods: 54 patients undergoing TKA were evaluated, measuring pre-op quadriceps strength, and utilizing the Oxford Knee Score for functionality. Post-op, we evaluated mobility using the Timed Up & Go, Elderly Mobility Scale, and Five Times Sit-to-Stand tests on POD 1 & 3/4. Pain levels, hospitalization, surgical duration, complications, and falls were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, over the age of 18, electively assigned for primary knee replacement surgery.
* ASA score 1-3

Exclusion Criteria:

* Revision surgery
* Patients suffering from chronic pain syndrome or chronic opioid use.
* Patients with previous neurological deficits in the lower extremities.
* A cognitive state that does not allow signing of consent or understanding simple instructions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Timed up & go test | first and fifth day after the surgery
  Total time to arise from chair, walk 3 m, turn around, return to chair and sit down. Two trials performed and the faster of the two is recorded to the nearest 10th of a second.
Change in Elderly mobility scale | first and fifth day after the surgery
  The EMS is a 20 point validated assessment tool for the assessment of frail elderly subjects. The EMS is measured on an ordinal scale of 0-20, when Scores under 10 - generally these patients are dependent in mobility manoeuvres; require help with basic ADL, such as transfers, toileting and dressing. Scores between 10 - 13 - generally these patients are borderline in terms of safe mobility and independence in ADL i.e. they require some help with some mobility manoeuvres.
  Scores over 14 - Generally these patients are able to perform mobility manoeuvres alone and safely and are independent in basic ADL.
Change in 5 times sit to stand test | first and fifth day after the surgery
  The score is the amount of time (to the nearest decimal in seconds) it takes a patient to transfer from a seated to a standing position and back to sitting five times.
Change in Numeric pain rating scale | up to five days
  An 11-point scale scored from 0 to 10: 0 = no pain, 10= the most intense pain imaginable
Chane in Quadriceps muscle strength | A 1 day before the surgery, first and fifth day after the surgery.
  muscle strength measure by dynamometer (N⋅m)

SECONDARY OUTCOMES:
Hospitalization duration | At discharge (assessed up to day 10)
  Number of days of hospitalization after the surgery- taken from the patient's file
Surgery duration | During the surgery
  minutes- taken from the patient's file
consumption of analgesics | At discharge (assessed up to day 10)
  taken from the patient's file
occurrence of falls | At discharge (assessed up to day 10)
  throughout the hospitalization- taken from the patient's file

OTHER OUTCOMES:
Oxford knee score questionnaire | A 1 day before the surgery
  The OKS is a patient self-completion PRO containing 12 questions on activities of daily living. It provides a single summed score which reflects the severity of problems that the respondent has with their knee. The OKS is scored 0-48 when Score 0-19 May indicate severe knee arthritis. Score 20-29 May indicate moderate to severe knee arthritis. Score 30-39 May indicate mild to moderate knee arthritis. Score 40-48 May indicate satisfactory joint function.

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shtarker, Dr, Principal Investigator — Head of the orthopedic department, Galilee medical center
Locations (1):
- Galilee medical center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kliger-Tendler M, Elboim-Gabyzon M, Bathish E, Shtarker H. Assessing Functional Outcomes and Pain Intensity Variations After Total Knee Arthroplasty: A Comparative Analysis of Pain Block Techniques. J Am Acad Orthop Surg Glob Res Rev. 2025 May 13;9(5):e24.00323. doi: 10.5435/JAAOSGlobal-D-24-00323. eCollection 2025 May 1. PMID 40388473